CLINICAL TRIAL: NCT01351168
Title: A Randomized, Controlled, Double-Blind, Cross-over Study of Zolpidem for Patients With Parkinson's Disease
Brief Title: Use of Zolpidem in Parkinson's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study not funded
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Leonard Verhagen Metman, MD, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZOL-PD
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; zolpidem
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; carbidopa, levodopa drug combination; Zolpidem; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: sugar pill
- Levodopa (Active Comparator)
  Interventions: Drug: Levodopa
- Zolpidam second dose (Experimental)
  Interventions: Drug: Zolpidem second dose
- Zolpidam first dose (Experimental)
  Interventions: Drug: Zolpidem first dose

INTERVENTIONS:
Drug: Levodopa — CD/LD 25/100, 2 tablets test dose based on subject's current CD/LD dosing; single randomized testing day
  Other Names: Sinemet
  Arms: Levodopa
Drug: Zolpidem first dose — Zolpidem will be given at 10 mg on randomized testing day. The randomization is such that the first dose of Zolpidem given to any subject will always be 10 mg
  Other Names: Ambien
  Arms: Zolpidam first dose
Drug: Zolpidem second dose — Zolpidem will be given at 7.5mg or 15 mg depending on the response from the first zolpidem dose.
  Other Names: Ambien
  Arms: Zolpidam second dose
Drug: sugar pill — a sugar pill (placebo) will all be given orally in identical capsules to the other study drugs
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
Levodopa treatment is associated with long-term complications. Dopamine deficiency is associated with abnormal activity in certain parts of the brain. Zolpidem may change this abnormal activity and, by doing so, may work in a different way than levodopa to help parkinsonism.

The working hypothesis for this aim is that ZLP is superior to placebo in acutely improving motor symptoms of PD. The investigators will conduct a randomized,controlled, double-blind, cross-over study in 40 patients with PD. Each patient will receive placebo, levodopa and 2 doses of ZLP in a randomized order on 4 different occasions, about one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have Idiopathic Parkinson's disease according to diagnostic criteria of the United Kingdom Parkinson's Disease Society Brain Bank.
* Subjects will be capable and willing to provide written informed consent prior to participation.
* Subjects will be ambulatory (in ON- and OFF-states) men and women, between the ages of 30 and 75 years.
* Subjects will be on levodopa therapy, with a good response and indisputable motor fluctuations.
* All other PD medications are allowed.
* Subjects will be on a stable regimen of PD medications for 2 weeks prior to screening.
* Subjects will be required to come with a caregiver who can accompany the subject to/from each study visit. Note: Subjects will not be allowed to drive home.
* Female subjects will be advised to use adequate birth control throughout the study as the effects of ZLP on the fetus are unknown. Adequate birth control methods include surgical sterilization, a partner who has had a vasectomy, oral contraceptives, condom plus spermicidal cream/jelly, cervical cap plus spermicidal cream/jelly, diaphragm plus spermicidal cream/jelly, or intrauterine device (in place for at least 3 months) plus spermicidal cream/jelly. Abstinence is considered an acceptable contraceptive regimen. If a subject becomes pregnant during the study, it is important that they contact the study physician immediately.

Exclusion Criteria:

* Neurodegenerative diseases.
* Tremor predominant PD, with a score of > 2 in more than one body part.
* Inability to tolerate being off levodopa for 12 hours.
* A score on the Montreal Cognitive Assessment (MoCA) of less than 26.
* Pregnancy or lactation.
* History of drug or alcohol abuse.
* Known or suspected sensitivity to the investigational study drugs.
* Other known medical or psychiatric condition that may compromise participation in the study or that judged by the site investigator could disqualify a subject from entering the study.
* Participation in another investigational drug study whereby they received experimental drug < 30 days prior to start of this study.
* Subjects who have undergone surgical procedures for PD but otherwise meet inclusion criteria will not be excluded a priori but evaluated on an individual basis.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
UPDRS | Subjects rated using the UPDRS at the Screening visit and then at each of the 4 study visits (1-2 weeks apart). During the study visits subjects will be rated every 30 minutes until they return to baseline.
  Unified Parkinson's Disease Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leo Verhagen, MD PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States